CLINICAL TRIAL: NCT01256814
Title: SystemCHANGE-HIV: A Pilot Study Exploring the Effect of a Systems-based Intervention to Increase Physical Activity, Sleep Behavior, and Mental Wellness
Brief Title: Study of SystemCHANGE-HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: Association of Nurses in AIDS Care (Other)
Responsible Party: Principal Investigator, Allison Webel, Instructor and Clinical Research Scholar, Case Western Reserve University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SystemCHANGE-HIV
Record Dates: First submitted 2010-12-08; First posted 2010-12-09 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: HIV
Keywords: HIV/AIDS; Adult; Behavioral Intervention; Sleep; Physical Activity
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behaviorial Intervention (Experimental): SystemCHANGE-HIV is a 10-week, small-group intervention that will promote behavior changes to improve the following: physical activity, sleep behaviors and mental wellness. S
  Interventions: Behavioral: SystemCHANGE-HIV
- Control (Active Comparator): The control group will receive the manual "Symptom Management Manual: Strategies for People Living with HIV/AIDS".
  Interventions: Behavioral: SystemCHANGE-HIV

INTERVENTIONS:
Behavioral: SystemCHANGE-HIV — SystemCHANGE, is based on social ecological theory and focuses on redesigning the family environment and daily routines that are linked to health behavior. This framework emphasizes context and specifies that change is best accomplished by: identifying a measurable goal, examining the system processes surrounding attainment of that goal, listing several ideas that may improve the system, engaging in a series of experiments to test the best ideas to improve the process, implementing the most successful ideas based on data from the experiments, and monitoring the system to maintain the gains. The SystemCHANGE-HIV intervention works to help participants make small environmental changes made in family daily routines that will eventually construct an environment.

SUMMARY:
The purpose of this study is to assess a new behavioral intervention to help how people living with HIV/AIDS practice self-management skills. Specifically, we want to see if a new educational intervention can improve physical activity, sleep, mental wellness and quality of life in HIV(Human Immunodeficiency Virus)-infected men and women. We hypothesize that those who are in the intervention group will practice more self-management skills than those in the control group.

DETAILED DESCRIPTION:
Sample: The study sample will include 40 HIV+ men and women. Inclusion criteria include: a documented HIV diagnosis; adult (18 years old or greater); and English speaking.

Design: The SystemCHANGE-HIV study will be a 15-week, randomized, two-group experimental design including a 10-week behavioral intervention. In the experimental group, one half of the participants (n=20) will receive the intervention; and in the control group, the other half of the participants will undergo usual care. Both the experimental and control group will complete the same psychometric instrument packet, three times, to give a comparison of self-management before and after intervention and at a four-week follow up visit. This packet includes information on medical history, demographics, HIV self-management,physical activity, social support, social capital, mental wellness, and quality of life.Additionally, all participants will wear an actigraph for seven consecutive days, at each data collection point, to assess sleep.

Analysis:Preliminary data analysis will include descriptive statistics and scatter plots to examine the distribution of each outcome at each time point, as well as each covariate of interest. Although our randomization scheme will ensure balance of baseline variables between the two arms (other than that due to chance alone), we will estimate the standardized magnitude of each baseline difference as well as the correlation between each baseline variable and each outcome of interest at 10 weeks or at 15 weeks to objectively determine baseline variables that will be needed to estimate the unbiased effect of the intervention on each outcome. The primary analysis will be based on intent to treat approach and will investigate the effect of the intervention on continuous outcomes at 10 weeks or 15 weeks. In particular, an Analysis of Covariance model will be used that adjusts for treatment arm and the baseline level of the outcome variable. Such a model will allow us to estimate the effect of the intervention on each outcome, adjusting for the baseline outcome.In addition, linear mixed models will be used to determine if the effect of the intervention on the outcome at 10 weeks differs from the effect of the intervention on the outcome at 15 weeks. If needed, all analyses will be repeated using an as-treated approach. All analyses will be performed using a two-sided significance of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* documented HIV diagnosis
* adult (21 years old or greater)
* English speaking

Exclusion Criteria:

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-01; Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Sleep quantity and quality | 15 weeks

SECONDARY OUTCOMES:
Physical Activity | 15 weeks
Mental Wellness | 15 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

REFERENCES:
- [Background] Lorig KR, Holman H. Self-management education: history, definition, outcomes, and mechanisms. Ann Behav Med. 2003 Aug;26(1):1-7. doi: 10.1207/S15324796ABM2601_01. PMID 12867348
- [Background] Beaglehole R, Epping-Jordan J, Patel V, Chopra M, Ebrahim S, Kidd M, Haines A. Improving the prevention and management of chronic disease in low-income and middle-income countries: a priority for primary health care. Lancet. 2008 Sep 13;372(9642):940-9. doi: 10.1016/S0140-6736(08)61404-X. PMID 18790317
- [Background] Burton NW, Haynes M, Wilson LA, Giles-Corti B, Oldenburg BF, Brown WJ, Giskes K, Turrell G. HABITAT: A longitudinal multilevel study of physical activity change in mid-aged adults. BMC Public Health. 2009 Mar 5;9:76. doi: 10.1186/1471-2458-9-76. PMID 19265552
- [Background] Glanz K, Bishop DB. The role of behavioral science theory in development and implementation of public health interventions. Annu Rev Public Health. 2010;31:399-418. doi: 10.1146/annurev.publhealth.012809.103604. PMID 20070207
- [Background] Kok G, Gottlieb NH, Commers M, Smerecnik C. The ecological approach in health promotion programs: a decade later. Am J Health Promot. 2008 Jul-Aug;22(6):437-42. doi: 10.4278/ajhp.22.6.437. PMID 18677885
- [Background] Jean-Louis G, Kripke DF, Mason WJ, Elliott JA, Youngstedt SD. Sleep estimation from wrist movement quantified by different actigraphic modalities. J Neurosci Methods. 2001 Feb 15;105(2):185-91. doi: 10.1016/s0165-0270(00)00364-2. PMID 11275275
- [Background] Moore SM, Charvat JM, Gordon NH, Pashkow F, Ribisl P, Roberts BL, Rocco M. Effects of a CHANGE intervention to increase exercise maintenance following cardiac events. Ann Behav Med. 2006 Feb;31(1):53-62. doi: 10.1207/s15324796abm3101_9. PMID 16472039
- [Background] Moore SM, Charvat JM. Using the CHANGE intervention to enhance long-term exercise. Nurs Clin North Am. 2002 Jun;37(2):273-83, vi-vii. doi: 10.1016/s0029-6465(01)00008-1. PMID 12389268